CLINICAL TRIAL: NCT02218021
Title: A Randomized, Double-Blind, Placebo- and Positive-Controlled, Crossover Study to Evaluate the Abuse Potential and Safety of Orally Administered Samidorphan in Non-Dependent Recreational Opioid Users
Brief Title: A Study of the Abuse Liability Potential of Samidorphan in Healthy, Non-Dependent, Recreational Opioid Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ALK33-012
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Volunteers
Keywords: Alkermes; ALKS 33; ALKS 5461; Samidorphan
MeSH Terms: interventions — 3-carboxamido-4-hydroxynaltrexone; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Samidorphan Dose 1 (Experimental)
  Interventions: Drug: Samidorphan
- Samidorphan Dose 2 (Experimental)
  Interventions: Drug: Samidorphan
- Samidorphan Dose 3 (Experimental)
  Interventions: Drug: Samidorphan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Oxycodone Dose 1 (Active Comparator)
  Interventions: Drug: Oxycodone
- Oxycodone Dose 2 (Active Comparator)
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Samidorphan
  Arms: Samidorphan Dose 1; Samidorphan Dose 2; Samidorphan Dose 3
Drug: Placebo
  Arms: Placebo
Drug: Oxycodone
  Arms: Oxycodone Dose 1; Oxycodone Dose 2

SUMMARY:
The purpose of this study is to evaluate the abuse potential and safety of samidorphan in healthy, non-dependent, adult, recreational opioid users.

ELIGIBILITY:
Inclusion Criteria:

* Be in good general physical health
* Body mass index of 18-34 kg/m2, inclusive with minimum weight of 50 kg
* Recreational opioid use experience for non-therapeutic purposes (at >/= 10 times in lifetime and >/= 1 in previous 3 months
* Agree to use an approved method of birth control for the duration of the study
* Additional criteria may apply

Exclusion Criteria:

* Currently pregnant or breastfeeding
* History of or current infection with hepatitis B virus, hepatitis C virus or HIV
* Current or history of any clinically significant medical or psychiatric condition
* Current or history of in the last 2 years of dependence on alcohol or any illicit drugs
* Have used any prescription or over-the-counter medication, including natural health products (with the exception of prescription birth control or hormonal replacements, acetaminophen, ibuprofen, or multivitamins) within 14 days
* Have a history of intolerance or hypersensitivity to opioid antagonists, opioid agonists or related drugs (eg, naltrexone, naloxone, oxycodone, morphine)
* Additional criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics: Abuse potential measured by visual analog scales (VAS) | Approximately 4 weeks

SECONDARY OUTCOMES:
Safety: Incidence of adverse events (AEs) | Approximately 5.5 weeks
Pharmacokinetics: Plasma concentrations of samidorphan and metabolite | Approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Pathak, MD, Study Director — Alkermes, Inc.
Locations (1):
- Alkermes Investigational Site, Overland Park, Kansas, United States